CLINICAL TRIAL: NCT02606747
Title: The Balance Control Mechanism of Diabetic Peripheral Neuropathy Patients
Brief Title: The Balance Control Mechanism of DPN Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Geheng Yuan (Other)
Responsible Party: Sponsor-Investigator, Geheng Yuan, Peking University first hospital, Peking University
Organization: Peking University (Other)
Other Study IDs: 11372013
Record Dates: First submitted 2015-04-09; First posted 2015-11-17 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Diabetic Neuropathy
Keywords: DPN; fall; fMRI; balance
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Diabetes mellitus with DPN: Aged from 40 to 80. Normal cognitive ability. Right handed. Able to walk without any other kinds of central nervous system disorder. Confirmed diabetes with DPN.
- Diabetes mellitus without DPN: Aged from 40 to 80. Normal cognitive ability. Right handed. Able to walk without any other kinds of central nervous system disorder. Confirmed diabetes without DPN.

INTERVENTIONS:
Other:  — routine blood sugar control

SUMMARY:
This study will evaluate the balance ability of DPN (diabetic peripheral neuropathy)patients, which will help us to understand the relationship between peripheral and central nervous system, in order to early diagnosis and prevent the fall in DPN patients.

DETAILED DESCRIPTION:
DPN is one of the most common complications of diabetes. The clinical manifestation of DPN contains sensory reduction, pain, muscle wastage and so on. Sensory and motor nervous are one of the most important factors in balance control, the reduction of balance ability will result in high risk of fall.

Most studies about DPN are focus on peripheral nervous, however, the central nervous system may also be involved in DPN patients. In this study, force platform, proprioception test and fMRI will be used to evaluate balance ability, proprioception and the brain function information of DPN patients, which will help to understand the relationship between peripheral and central nervous system.

ELIGIBILITY:
Inclusion Criteria:

* diabetics
* normal cognitive ability
* walk normally
* normal vision

Exclusion Criteria:

* other nervous system disease, foot ulcer

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetics
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Scale | through study completion, an average of 6 months; Berg Balance Scale assessment
  In Berg Balance Scale, 14-item scale designed to measure balance of the adult in a clinical setting, including sitting to standing, standing unsupported, sitting unsupported, standing to sitting, transfers, standing with eyes closed, standing with feet together, reaching forward with outstretched arm, retrieving object from floor, turning to look behind, turning 360 degrees, placing alternate foot on stool, standing with one foot in front and standing on one foot. For each item, a five-point scale ranging from 0-4 was recorded. "0" indicates the lowest level of function and "4" the highest level of function. Total Score = 56.
Brain complexity and connectivity | through study completion, an average of 6 months; brain complexity and connectivity assessment
  Brain complexity and connectivity was assessed by fMRI (functional magnetic resonance imaging).
  For each patient, an 8 minutes resting state fMRI signal was recorded. Brain complexity and connectivity was calculated from fMRI signal. By using AAL (automated anatomical labeling) template, the brain was separated into 90 regions. The complexity of each brain region was calculated and range from 50 to 100. "50" indicates the lowest complexity and "100" indicates the highest complexity. The connectivity between each region was also calculated and range from 0 to 1. "0" indicates the weakest connectivity and "1" indicates the strongest connectivity.
  The brain complexity and connectivity in both DPN group and diabetics without DPN group could help us to explore the brain differences between two groups.
Timed up and go | through study completion, an average of 6 months; timed up and go assessment
  Timed up and go test was to assess the walk speed of patients. In timed up and go test, the patient sit on a standard armchair and used regular footwear. The patient walk to a line that is 3 meters away, turn around at the line, walk back to the chair, and sit down. The test ends when the patient's buttocks touch the seat. Patients were instructed to use a comfortable and safe walking speed. A stopwatch was used to time the test (in seconds).
Foot sole tactile threshold | through study completion, an average of 6 months; foot sole tactile threshold assessment
  The foot sole tactile threshold test was to assess the vibration sensation of patients. In foot sole tactile threshold test, the patient was instructed to stand on a pair of vibration insoles. The vibration amplitude was adjusted by experimenter until the patient cannot aware the vibration. The vibration threshold of each foot was recorded from 1 to 100. "1" indicates the weakest vibration and "100" indicates the strongest vibration.

CONTACTS AND LOCATIONS:
Overall Officials: Jue Zhang, Ph. D, Study Chair — PKU
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China